CLINICAL TRIAL: NCT00503347
Title: A Phase Ib Open-Label, Escalating Repeat-Dose Trial of Bavituximab (Chimeric Anti-Phosphatidylserine Monoclonal Antibody) in Patients Co-Infected With Chronic Hepatitis C Virus and Human Immunodeficiency Virus
Brief Title: Bavituximab Repeat-Dose Trial in Patients Co-Infected With Chronic Hepatitis C Virus and Human Immunodeficiency Virus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peregrine Pharmaceuticals (Industry)
Responsible Party: Jill Capps / Clinical Program Manager, Peregrine Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPHM 0603
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Hepatitis C Virus; Hiv Infections
Keywords: coinfection with chronic hepatitis C virus and HIV; Treatment Naive
MeSH Terms: conditions — Hepatitis C; HIV Infections | interventions — bavituximab

ARMS (4):
- 1 (Experimental): 0.3 mg/kg
  Interventions: Drug: bavituximab
- 2 (Experimental): 1 mg/kg
  Interventions: Drug: bavituximab
- 3 (Experimental): 3 mg/kg
  Interventions: Drug: bavituximab
- 4 (Experimental): 6 mg/kg
  Interventions: Drug: bavituximab

INTERVENTIONS:
Drug: bavituximab — The study drug is a sterile solution administered intravenously weekly for 8 weeks. Each cohort is given 0.3, 1, 3, or 6 mg/kg of bavituximab.

SUMMARY:
This trial is designed to assess the safety, tolerability, pharmacokinetics and viral kinetics after multiple infusions of bavituximab in patients co-infected with HCV and HIV.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the safety and tolerability of bavituximab administered as multiple intravenous (IV) infusions to patients co-infected with HCV and HIV
* To characterize the pharmacokinetic profile and viral kinetics after multiple intravenous infusions of bavituximab to patients infected with HCV and HIV
* To define the maximum tolerated dose (MTD) and/or maximum effective dose (MED) of bavituximab administered as multiple infusions to patients infected with chronic HCV infection and HIV

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been obtained
* Adults 18 years of age or older
* HIV infection documented by detectable HIV RNA PCR
* Absolute CD4+ > 300 cells/mm3
* Chronic hepatitis C infection based on history and detectable serum HCV RNA
* Serum alanine aminotransferase (ALT) above normal limits and/or historical biopsy consistent with hepatitis C
* Complete blood counts within normal limits
* Normal renal function (serum creatinine within normal limits)
* PT/INR and aPTT within normal limits
* All patients of reproductive potential must agree to use an approved form of barrier contraception or agree not to become pregnant while taking study medications and for 30 days after study completion. Female patients must have a negative serum pregnancy test at prestudy (not applicable to patients with bilateral oophorectomy and/or hysterectomy or to those patients who are postmenopausal)

Exclusion Criteria:

* HCV or HIV antiviral therapy within 4 weeks of Day 0
* Prior exposure to any chimeric antibody
* Any other cause of liver disease other than chronic hepatitis C, such as autoimmune or alcoholic liver disease.
* Decompensated clinical liver disease, including a history of prolonged clotting times, hypoalbuminemia, encephalopathy, treatment for elevated ammonia levels, or ascites
* Any evidence of clinically significant bleeding defined as gross hematuria, hemoptysis, or gastrointestinal bleeding
* Known history of bleeding diathesis or coagulopathy (e.g., von Willebrand Disease or Hemophilia)
* Any history of thromboembolic events [e.g., deep vein thrombosis (DVT) or pulmonary thromboembolism (PE)]. A history of including central venous catheter-related thrombosis is acceptable if there is documentation of resolution at least 12 months prior to enrollment.
* Concurrent therapy with oral or parenteral anticoagulants
* Concurrent hormone therapy (i.e., estrogen contraceptives, hormone replacement, anti-estrogen)
* Investigational therapy within 4 weeks of Day 0
* Major surgery within 4 weeks of Day 0
* Pregnant or nursing women
* Uncontrolled intercurrent disease (e.g., diabetes, hypertension, thyroid disease)
* Any history of angina pectoris, coronary artery disease or cerebrovascular accident, or transient ischemic attack
* A history of any condition requiring anti-platelet therapy with the exception of general cardiovascular prophylaxis with aspirin
* A history of any condition requiring treatment (past or current) with coumarin-type agents
* Cardiac arrhythmia requiring medical therapy
* Serious non-healing wound (including wound healing by secondary intention, ulcer, or bone fracture)
* Requirement for chronic daily treatment with NSAIDs, antiplatelet drugs (e.g., phosphodiesterase inhibitors, adenosine diphosphate receptor antagonists), or steroids
* Cancer, autoimmune disease or any disease or concurrent therapy known to cause significant alteration in immunologic function. Corticosteroids administered as pre-treatment, or to treat an adverse event, are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-07; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
• Adverse events • Laboratory evaluations • Human anti-chimeric antibody • Pharmacokinetic analysis

SECONDARY OUTCOMES:
Blood levels of HCV RNA and HIV RNA (PCR)

CONTACTS AND LOCATIONS:
Overall Officials: Jihad Slim, MD, Principal Investigator — Saint Michael's Medical Center; Mark S. Sulkowski, MD, Principal Investigator — Johns Hopkins University, Center for Viral Hepatitis; Jorge Rodriguez, MD, Principal Investigator — Orange Coast Medical Center; Nicholaos C. Bellos, MD, Principal Investigator — Southwest Infectious Disease Associates; Lydie Hazan, MD, Principal Investigator — Impact Clinical Trials; Melaine Thompson, MD, Principal Investigator — AIDS Research Consortium of Atlanta (ARCA)
Locations (6):
- United States (6):
  - Impact Clinical Research, Los Angeles, California
  - Orange Coast Medical Center, Newport Beach, California
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Johns Hopkins University, Center for Viral Hepatitis, Baltimore, Maryland
  - Saint Michael's Medical Center, Newark, New Jersey
  - Southwest Infectious Disease Associates, Dallas, Texas